CLINICAL TRIAL: NCT06980324
Title: Effect of Integrated Neuromuscular Inhibition Technique on Iliotibial Band Friction Syndrome
Brief Title: Neuromuscular Inhibition Technique on Iliotibial Band Friction Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Tarek Farouk, Basic science physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/004885
Record Dates: First submitted 2025-03-23; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-10

CONDITIONS: Iliotibial Band Syndrome
Keywords: integrated neuromuscular inhibition technique; iliotibial band friction syndrome; muscle energy technique; ischemic compression; positional release
MeSH Terms: conditions — Iliotibial Band Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Experimental)
  Interventions: Other: conventional physical therapy treatment
- Interventional group (Experimental)
  Interventions: Other: integrated neuromuscular inhibition technique

INTERVENTIONS:
Other: integrated neuromuscular inhibition technique — integrated neuromuscular inhibition technique consists of:
  * ischemic compression
  * Positional release
  * Muscle energy technique
  Arms: Interventional group
Other: conventional physical therapy treatment — Conventional physical therapy treatment:
  * Ultrasound
  * Hotpacks
  * Iliotibial band stretching
  * Static quadriceps and hamstring exercises
  Arms: control group

SUMMARY:
The goal of this clinical trial is to find the effect of integrated neuromuscular inhibition technique for iliotibial band in iliotibial band friction syndrome on pain intensity level, pressure pain threshold, knee range of motion, knee function and knee angle . The main questions it aims to answer are:

* Is there an effect of integrated neuromuscular inhibition technique for iliotibial band on pain intensity level in iliotibial band friction syndrome?
* Is there an effect of integrated neuromuscular inhibition technique for iliotibial band on pressure pain threshold in iliotibial band friction syndrome?
* Is there an effect of integrated neuromuscular inhibition technique for iliotibial band on knee range of motion in iliotibial band friction syndrome?
* Is there an effect of integrated neuromuscular inhibition technique for iliotibial band on knee function in iliotibial friction syndrome? Is there an effect of integrated neuromuscular inhibition technique for iliotibial band on knee angle in iliotibial band friction syndrome?

Researchers will compare integrated neuromuscular inhibition technique to conventional physiotherapy to see if integrated neuromuscular inhibition technique works to treat iliotibial band syndrome.

Participants will:

* Take sessions for 2 weeks
* Visit the department 3 times per week

ELIGIBILITY:
Inclusion Criteria:

* Body mass index from 25-30 kg/m2
* Both males and females will be included their age from 30-50.
* The subjects that will be included in the study will be referred from orthopeadic physician with iliotibial band friction syndrome with these signs and symptoms
* local tenderness of the lateral knee inferior to the epicondyle and superior to the joint line
* Pain with ITBS can be reported anywhere along the iliotibial (IT) band from the lateral thigh to the lateral femoral condyle and Gerdy's tubercle.
* Pain is most intense at approximately 30 degrees of knee.
* A sharp, burning pain when the practitioner presses on the lateral epicondyle during knee flexion and extension associated with one of these cases:
* Tibiofermoral knee pain.
* Patellofemoral knee pain.
* osteoarthritis with medial knee joint pain
* Lateral patellar pressure syndrome.
* Medial meniscus degeneration.
* Excessive lateral pressure syndrome

Exclusion Criteria:

* Traumatic injury to the knee joint within 6 months.
* Surgical procedure on the affected knee within the last 12 months.
* Meniscus injury
* knee ligaments injury
* Malignancies, tumors or infections associated with the knee joint.
* Impaired thermal sensation over the knee.
* Subject with psychiatric disorder.
* Peripheral vascular disease.
* Severe joint deformity.
* Current back or ankle pain.
* Rheumatoid arthritis.
* Lower extremity fracture.
* Neurological defecit or movement disorder.
* Athletes.
* Menopause
* Pregnancy
* Auto immune disease
* Chronic disease (Diabetes mellitus and Hypertension)

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | after 2 weeks
  The Visual Analogue Scale (VAS) was used to evaluate pain severity. It is a self-reported pain measurement scale, consisting of a horizontal or vertical line, usually 10 cm long. The extremes of the line are labeled as no pain and worst pain. Each subject was asked to mark the point on the line that exactly corresponded to his/her pain
lower extremity function | after 2 weeks
  Lower extremity functional scale (LEFS):
  LEFS is a questionnaire containing 20 items assessing the lower extremity function based on the intensity of the related activities' performance. This scoring system is designed based on the five-score Likert scale ranging from zero as the worst condition to four as without bothersome. This scale scores from zero to eighty and the higher score represent a better condition. LEFS-Arabic version will be used to quantify activity limitation in Arabic-speaking individuals with lower extremity musculoskeletal disorders
Knee range of motion | after 2 weeks
  Digital goniometer:
  A goniometer is a device that measures an angle or permits the rotation of an object to a definite position .To measure knee joint ROM goniometer was lined up with the lateral side of femur with the proximal arm between trochanter major and the middle of the lateral joint space of the knee and the distal arm between the middle of the lateral joint space of the knee and the lateral malleoli

SECONDARY OUTCOMES:
pressure pain threshold | after 2 weeks
  The pressure algometer was applied three times at each of the three marked points. Each application of the pressure algometer was stopped when the participant perceived a change in sensation from pressure to pain at the measurement point. Using a mechanical pressure Fischer algometer .
  Pressure was increased with a speed (1kg/cm2). Steady and perpendicular to the identified trigger point, subjects were instructed to say "now" when they first began to feel change of pressure to either discomfort or pain. The mean of 3 trials over each point was calculated. It is important to place the tip of the algometer precisely on the MTrP region to avoid any major difference in readings among the consecutive measurements of the same MTrP.
knee angle | after 2 weeks
  Kinovea is one of the most commonly used applications. Kinovea is a free 2D motion analysis software for computers that can be used to measure kinematic parameters.
  Subjects were required to stand and relaxed lower limbs, with feet forward and shoulder-width apart. The camera was set 3 m from the subject .
  The vertical axis of the camera was aligned with the midpoint between the lower limbs of the participant. The image was zoomed to the closest capture, where the stickers could be clearly visible, and always set in the same position.

CONTACTS AND LOCATIONS:
Overall Officials: AMIR MO Saleh, Professor of Physical Therapy, Study Chair — Cairo University; Doaa RA Elazab, Assistant professor, Study Director — Cairo University; Hassan HU Ahmed, Orthopedic Surgery Professor, Study Director — Faculty of Medicine Banha University; Esraa TA Farouk, Physical therapist, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaughan, Brett (external link) and McLaughlin, Patrick (2014) Immediate changes in pressure pain threshold in the Iliotibial band using a myofascial (foam) roller. International Journal of Therapy and Rehabilitation, 21 (12). 569 - 574. ISSN 1741-1645
- [Background] Zimmermann SM, Njagulj V, Fritz B, Fucentese SF, Sutter R, Pfirrmann CWA. The Accessory Iliotibial Band-Meniscal Ligament of the Knee: Association With Lesions of the Lateral Meniscus. AJR Am J Roentgenol. 2019 Oct;213(4):912-917. doi: 10.2214/AJR.18.21071. Epub 2019 Jun 25. PMID 31237768
- [Background] Zhang DH, Wu ZQ, Zuo XC, Li JW, Huang CL. Diagnosis and treatment of excessive lateral pressure syndrome of the patellofemoral joint caused by military training. Orthop Surg. 2011 Feb;3(1):35-9. doi: 10.1111/j.1757-7861.2010.00116.x. PMID 22009978
- [Background] Whelton H, Harrington J, Crowley E, Kelleher V, Cronin M, Perry IJ. Prevalence of overweight and obesity on the island of Ireland: results from the North South Survey of Children's Height, Weight and Body Mass Index, 2002. BMC Public Health. 2007 Jul 31;7:187. doi: 10.1186/1471-2458-7-187. PMID 17672893
- [Background] Walsh TP, Arnold JB, Evans AM, Yaxley A, Damarell RA, Shanahan EM. The association between body fat and musculoskeletal pain: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2018 Jul 18;19(1):233. doi: 10.1186/s12891-018-2137-0. PMID 30021590
- [Background] Kang SY, Choung SD, Park JH, Jeon HS, Kwon OY. The relationship between length of the iliotibial band and patellar position in Asians. Knee. 2014 Dec;21(6):1135-8. doi: 10.1016/j.knee.2014.09.005. Epub 2014 Oct 12. PMID 25311516
- [Background] Macfarlane GJ, de Silva V, Jones GT. The relationship between body mass index across the life course and knee pain in adulthood: results from the 1958 birth cohort study. Rheumatology (Oxford). 2011 Dec;50(12):2251-6. doi: 10.1093/rheumatology/ker276. Epub 2011 Oct 8. PMID 21984765
- [Background] Vasilevska V, Szeimies U, Stabler A. Magnetic resonance imaging signs of iliotibial band friction in patients with isolated medial compartment osteoarthritis of the knee. Skeletal Radiol. 2009 Sep;38(9):871-5. doi: 10.1007/s00256-009-0704-z. Epub 2009 May 30. PMID 19484234
- [Background] Svensson M, Lind V, Lofgren Harringe M. Measurement of knee joint range of motion with a digital goniometer: A reliability study. Physiother Res Int. 2019 Apr;24(2):e1765. doi: 10.1002/pri.1765. Epub 2018 Dec 27. PMID 30589162
- [Background] Strauss EJ, Kim S, Calcei JG, Park D. Iliotibial band syndrome: evaluation and management. J Am Acad Orthop Surg. 2011 Dec;19(12):728-36. doi: 10.5435/00124635-201112000-00003. PMID 22134205
- [Background] Sorour AS, Ayoub AS, Abd El Aziz EM. Effectiveness of acupressure versus isometric exercise on pain, stiffness, and physical function in knee osteoarthritis female patients. J Adv Res. 2014 Mar;5(2):193-200. doi: 10.1016/j.jare.2013.02.003. Epub 2013 Apr 8. PMID 25685487
- [Background] Bassiouni H, Aly H, Zaky K, Abaza N, Bardin T. Probing The Relation Between Vitamin D Deficiency and Progression of Medial Femoro-tibial Osteoarthitis of the Knee. Curr Rheumatol Rev. 2017;13(1):65-71. doi: 10.2174/1573397112666160404124532. PMID 27041085
- [Background] Saadat Z, Hemmati L, Pirouzi S, Ataollahi M, Ali-Mohammadi F. Effects of Integrated Neuromuscular Inhibition Technique on pain threshold and pain intensity in patients with upper trapezius trigger points. J Bodyw Mov Ther. 2018 Oct;22(4):937-940. doi: 10.1016/j.jbmt.2018.01.002. Epub 2018 Jan 17. PMID 30368338
- [Background] Rupareliya JD, Donga S, Gandhi AJ. Management of Vandhyatva w.s.r. to thin endometrium through Ayurveda- A single arm open labelled pilot clinical trial. Ayu. 2021 Oct-Dec;42(4):156-163. doi: 10.4103/ayu.ayu_132_21. Epub 2023 May 17. PMID 37347080
- [Background] Noori SA, Rasheed A, Aiyer R, Jung B, Bansal N, Chang KV, Ottestad E, Gulati A. Therapeutic Ultrasound for Pain Management in Chronic Low Back Pain and Chronic Neck Pain: A Systematic Review. Pain Med. 2020 Nov 7;21(7):1482-1493. doi: 10.1093/pm/pny287. PMID 30649460
- [Background] Dobec-Meic B, Pikija S, Cvetko D, Trkulja V, Pazanin L, Kudelic N, Rotim K, Pavlicek I, Kostanjevec AR. Intracranial tumors in adult population of the Varazdin County (Croatia) 1996-2004: a population-based retrospective incidence study. J Neurooncol. 2006 Jul;78(3):303-10. doi: 10.1007/s11060-005-9100-2. Epub 2006 Apr 6. PMID 16598428
- [Background] Koh RG, Paul TM, Nesovic K, West D, Kumbhare D, Wilson RD. Reliability and minimal detectable difference of pressure pain thresholds in a pain-free population. Br J Pain. 2023 Jun;17(3):239-243. doi: 10.1177/20494637221147185. Epub 2022 Dec 23. PMID 37342397
- [Background] Kinser AM, Sands WA, Stone MH. Reliability and validity of a pressure algometer. J Strength Cond Res. 2009 Jan;23(1):312-4. doi: 10.1519/jsc.0b013e31818f051c. PMID 19130648
- [Background] Imamura M, Alfieri FM, Filippo TR, Battistella LR. Pressure pain thresholds in patients with chronic nonspecific low back pain. J Back Musculoskelet Rehabil. 2016 Apr 27;29(2):327-336. doi: 10.3233/BMR-150636. PMID 26406214
- [Background] Hutchinson LA, Lichtwark GA, Willy RW, Kelly LA. The Iliotibial Band: A Complex Structure with Versatile Functions. Sports Med. 2022 May;52(5):995-1008. doi: 10.1007/s40279-021-01634-3. Epub 2022 Jan 24. PMID 35072941
- [Background] Hamstra-Wright KL, Jones MW, Courtney CA, Maiguel D, Ferber R. Effects of iliotibial band syndrome on pain sensitivity and gait kinematics in female runners: A preliminary study. Clin Biomech (Bristol). 2020 Jun;76:105017. doi: 10.1016/j.clinbiomech.2020.105017. Epub 2020 Apr 30. PMID 32388078
- [Background] Lashien SA, Abdelnaeem AO, Gomaa EF. Effect of hip abductors training on pelvic drop and knee valgus in runners with medial tibial stress syndrome: a randomized controlled trial. J Orthop Surg Res. 2024 Oct 29;19(1):700. doi: 10.1186/s13018-024-05139-3. PMID 39468623
- [Background] Ferber R, Noehren B, Hamill J, Davis IS. Competitive female runners with a history of iliotibial band syndrome demonstrate atypical hip and knee kinematics. J Orthop Sports Phys Ther. 2010 Feb;40(2):52-8. doi: 10.2519/jospt.2010.3028. PMID 20118523
- [Background] Farrokhi S, Chen YF, Piva SR, Fitzgerald GK, Jeong JH, Kwoh CK. The Influence of Knee Pain Location on Symptoms, Functional Status, and Knee-related Quality of Life in Older Adults With Chronic Knee Pain: Data From the Osteoarthritis Initiative. Clin J Pain. 2016 Jun;32(6):463-70. doi: 10.1097/AJP.0000000000000291. PMID 26308705
- [Background] Farasyn A. (2007) Pressure pain algometry in patients with non-specific low back pain. Faculty of Physical Education and Physiotherapy Department of Human Physiology & Sports Medicine
- [Background] Evans P. The postural function of the iliotibial tract. Ann R Coll Surg Engl. 1979 Jul;61(4):271-80. PMID 475270
- [Background] Dixit, M., Samal, S., & Ramteke, SEfficacy of Maitland Mobilization and Myofascial Trigger Point Release in Patients of Osteoarthritis of Knee. Indian Journal of Public Health Research & Development, (2020), 11(5), 705-710.
- [Background] Dekkers JC, van Wier MF, Hendriksen IJ, Twisk JW, van Mechelen W. Accuracy of self-reported body weight, height and waist circumference in a Dutch overweight working population. BMC Med Res Methodol. 2008 Oct 28;8:69. doi: 10.1186/1471-2288-8-69. PMID 18957077
- [Background] Danazumi MS, Yakasai AM, Ibrahim AA, Shehu UT, Ibrahim SU. Effect of integrated neuromuscular inhibition technique compared with positional release technique in the management of piriformis syndrome. J Osteopath Med. 2021 May 31;121(8):693-703. doi: 10.1515/jom-2020-0327. PMID 34049428
- [Background] Crossley KM, Callaghan MJ, van Linschoten R. Patellofemoral pain. Br J Sports Med. 2016 Feb;50(4):247-50. doi: 10.1136/bjsports-2015-h3939rep. PMID 26834209
- [Background] Chitale N Jr, Patil DS, Phansopkar P. Integrated Neuromuscular Inhibition Technique Versus Mulligan Mobilization on Functional Disability in Subjects With Nonspecific Low Back Pain: A Comparative Study. Cureus. 2022 Oct 13;14(10):e30253. doi: 10.7759/cureus.30253. eCollection 2022 Oct. PMID 36381847
- [Background] Chevalier A, Van Overmeire A, Vermue H, Pringels L, Herregodts S, Victor J, Loccufier M. Effect of iliotibial band and gastrocnemius activation on knee kinematics. Knee. 2023 Jan;40:238-244. doi: 10.1016/j.knee.2022.11.025. Epub 2022 Dec 13. PMID 36521416
- [Background] Bose K, Kanagasuntheram R, Osman MB. Vastus medialis oblique: an anatomic and physiologic study. Orthopedics. 1980 Sep 1;3(9):880-3. doi: 10.3928/0147-7447-19800901-12. PMID 24822568
- [Background] Begum M.R. (2019) Validity and reliability of visual analogue scale (vas) for pain measurement. Journal of Medical Case Reports and Reviews 2.
- [Background] Al-Najjar, H. M. M., Mohammed, A. H., & Mosaad, D. M. Effect of ice massage with integrated neuromuscular inhibition technique on pain and function in subjects with mechanical neck pain: randomized controlled trial. Bulletin of Faculty of Physical Therapy, (2020), 25, 1-7
- [Background] Alnahdi AH, Alrashid GI, Alkhaldi HA, Aldali AZ. Cross-cultural adaptation, validity and reliability of the Arabic version of the Lower Extremity Functional Scale. Disabil Rehabil. 2016;38(9):897-904. doi: 10.3109/09638288.2015.1066452. Epub 2015 Jul 17. PMID 26186622
- [Background] Ali Ismail AM, Abd El-Azeim AS, El-Sayed Felaya EE. Integrated neuromuscular inhibition technique versus spray and stretch technique in neck pain patients with upper trapezius trigger points: a randomized clinical trial. J Man Manip Ther. 2024 Apr;32(2):141-149. doi: 10.1080/10669817.2023.2192899. Epub 2023 Mar 23. PMID 36951194
- [Background] Abaza SE. The dilemma of knee osteoarthritis and iliotibial band syndrome. MOJ Orthop Rheumatol. 2015,2(4):145-146.